CLINICAL TRIAL: NCT02710760
Title: Translating Adoption of Improved Varieties Into Nutritional Impact for Young Children: An RCT Exploring Strategies to Increase Consumption of Quality Protein Maize in Ethiopia
Brief Title: Translating Adoption of Improved Varieties Into Nutritional Impact
Acronym: QPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: CIMMYT International Maize and Wheat Improvement Center (Unknown); Ethiopian Public Health Institute (Other Government); Agricultural Technology Adoption Initiative (Unknown)
Responsible Party: Principal Investigator, Jessica Cohen, Assistant Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB14-3255
Record Dates: First submitted 2016-02-29; First posted 2016-03-17 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Malnutrition
Keywords: Biomarkers; Child Nutrition Sciences; Economics, Behavioral
MeSH Terms: conditions — Malnutrition; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Households in the control group receive no special treatment.
- Adoption Encouragement Treatment (Experimental): Households in the Adoption Encouragement Treatment group were visited between March and April 2015 and offered "child nutrition focused" adoption encouragement. Both the male household head and the primary female caregiver were invited to attend these meetings (though the household head is the primary target), where the nutritional benefits of Quality Protein Maize (QPM) adoption for children were emphasized along with the agronomic properties. In addition, the fact that only small amounts of QPM are necessary to nourish children was highlighted and small seed bag sizes were offered. During the adoption encouragement visit, we offered the option to order up to three 2 kg bags of QPM for free.
  Interventions: Other: Adoption Encouragement Treatment
- Consumption Encouragement Treatment (Experimental): In addition to receiving the Adoption Encouragement Treatment, households in the Consumption Encouragement Treatment group received additional information, targeted to the caregiver, and tools for separating Quality Protein Maize and targeting it to young children in the household in August 2015. They will additionally receive further guidance in February 2016.
  Interventions: Other: Adoption Encouragement Treatment; Other: Consumption Encouragement Treatment

INTERVENTIONS:
Other: Adoption Encouragement Treatment — Households in the Adoption Encouragement Treatment received child nutrition focused guidance on the nutritional and agronomic benefits of Quality Protein Maize (QPM) adoption, and the opportunity to order up to 6 kg of QPM seed to plant in their own fields.
  Arms: Adoption Encouragement Treatment; Consumption Encouragement Treatment
Other: Consumption Encouragement Treatment — Households in the Consumption Encouragement Treatment received the same guidance as households in the Adoption Encouragement Treatment, as well as additional guidance on the importance of specifically targeting foods made with QPM to young children and tools to help households keep the grain separate and remember to feed QPM-based foods to the young children.
  Arms: Consumption Encouragement Treatment

SUMMARY:
The purposes of this study are (1) to determine whether child nutrition-focused adoption encouragement messages focused on Quality Protein Maize (QPM) and the availability of small quantities of QPM seed can be effective at increasing QPM adoption and health outcomes for young children, and (2) to determine whether consumption encouragement messages and techniques (e.g., containers for earmarking) can be effective at increasing QPM targeting to and health outcomes for young children.

ELIGIBILITY:
Inclusion Criteria:

Households with at least one child in the 6-35 month age range in August 2015, who had at least one household member attend a field day demonstrating Quality Protein Maize, and who provided informed consent for participation and data collection were eligible for inclusion.

Exclusion Criteria:

Households in the study areas that do not have a member who attends a field day demonstrating Quality Protein Maize or who do not have a child in the appropriate age range are excluded from the study. Furthermore, households where the mother or children did not intend on staying in the region for the study duration (until the completion of the endline survey) were excluded from the study. Finally, we excluded participants who do not have access to land for crop cultivation.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 978 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Consumption of any QPM by the index child in the last 24 hours | 6-7 months
Amount of QPM consumed by the index child in the last 24 hours | 6-7 months
Index child's proportion of total maize consumption that was QPM in the last 24 hours | 6-7 months
Consumption of any QPM by the index child in the last week | 6-7 months
Number of days in the last week that the index child ate any QPM | 6-7 months
Number of days in the last week that caregiver cooked a QPM-based food that was primarily for target children | 6-7 months
Height-for-age Z-score of index child | 6-7 months
Weight-for-height Z-score of index child | 6-7 months
Weight-for-age Z-score of index child | 6-7 months
Mid-upper arm circumference-for-age Z-score of index child | 6-7 months
Insulin-like growth factor I (continuous measurement) | 6-7 months
Amount of QPM reserved for home consumption | 6-7 months
Hectares of QPM planted | 6-7 months
Serum transthyretin | 6-7 months
Consumption of any QPM by the index child in the last 24 hours | 10-11 months
Amount of QPM consumed by the index child in the last 24 hours | 10-11 months
Index child's proportion of total maize consumption that was QPM in the last 24 hours | 10-11 months
Consumption of any QPM by the index child in the last week | 10-11 months
Number of days in the last week that the index child ate any QPM | 10-11 months
Number of days in the last week that caregiver cooked a QPM-based food that was primarily for target children | 10-11 months
Height-for-age Z-score of index child | 10-11 months
Weight-for-height Z-score of index child | 10-11 months
Weight-for-age Z-score of index child | 10-11 months
Mid-upper arm circumference-for-age Z-score of index child | 10-11 months
Amount of QPM reserved for home consumption | 10-11 months
Change in Height-for-age Z-score of index child | 6-7 months
Change in Height-for-age Z-score of index child | 10-11 months
Change in Weight-for-height Z-score of index child | 6-7 months
Change in Weight-for-height Z-score of index child | 10-11 months
Change in Mid-upper arm circumference-for-age Z-score of index child | 6-7 months
Change in Mid-upper arm circumference-for-age Z-score of index child | 10-11 months
Change in Weight-for-age Z-score of index child | 6-7 months
Change in Weight-for-age Z-score of index child | 10-11 months

SECONDARY OUTCOMES:
Serum lysine | 6-7 months
Serum tryptophan | 6-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cohen, PhD, Principal Investigator — Harvard Chan School of Public Health

IPD SHARING:
Plan to Share IPD: Yes
We will share completely deidentified data upon request after primary analyses have been been completed.

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Victora CG, Adair L, Fall C, Hallal PC, Martorell R, Richter L, Sachdev HS; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: consequences for adult health and human capital. Lancet. 2008 Jan 26;371(9609):340-57. doi: 10.1016/S0140-6736(07)61692-4. PMID 18206223
- [Background] Ruel MT, Alderman H; Maternal and Child Nutrition Study Group. Nutrition-sensitive interventions and programmes: how can they help to accelerate progress in improving maternal and child nutrition? Lancet. 2013 Aug 10;382(9891):536-51. doi: 10.1016/S0140-6736(13)60843-0. Epub 2013 Jun 6. PMID 23746780
- [Background] Masset E, Haddad L, Cornelius A, Isaza-Castro J. Effectiveness of agricultural interventions that aim to improve nutritional status of children: systematic review. BMJ. 2012 Jan 17;344:d8222. doi: 10.1136/bmj.d8222. PMID 22251864
- [Background] Girard AW, Self JL, McAuliffe C, Olude O. The effects of household food production strategies on the health and nutrition outcomes of women and young children: a systematic review. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:205-22. doi: 10.1111/j.1365-3016.2012.01282.x. PMID 22742612
- [Background] Ghosh S, Suri D, Uauy R. Assessment of protein adequacy in developing countries: quality matters. Br J Nutr. 2012 Aug;108 Suppl 2:S77-87. doi: 10.1017/S0007114512002577. PMID 23107551
- [Derived] Donato K, McConnell M, Han D, Gunaratna NS, Tessema M, De Groote H, Cohen J. Behavioural insights to support increased consumption of quality protein maize by young children: a cluster randomised trial in Ethiopia. BMJ Glob Health. 2020 Dec;5(12):e002705. doi: 10.1136/bmjgh-2020-002705. PMID 33355261